CLINICAL TRIAL: NCT00811538
Title: Swiss Intravenous and Intra-arterial Thrombolysis for Treatment of Acute Ischemic Stroke Registry (SWISS)
Brief Title: Swiss Intravenous and Intra-arterial Thrombolysis for Treatment of Acute Ischemic Stroke Registry
Acronym: SWISS
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Swiss Heart Foundation (Other); University of Zurich (Other); University Hospital, Basel, Switzerland (Other); University Hospital, Geneva (Other); University of Lausanne Hospitals (Other); Kantonsspital Aarau (Other); Cantonal Hospital of St. Gallen (Other); Triemli Hospital (Other)
Responsible Party: PD Dr. Marcel Arnold, Oberarzt, Dep. of Neurology, Bern University Hospital
Other Study IDs: 233/07; 1446; KEK 233/07 (Other: Ethics Committee)
Record Dates: First submitted 2008-12-18; First posted 2008-12-19 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Ischemic Stroke
Keywords: ischemic stroke; endovascular treatment; Thrombolysis; outcome
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1 1 (Liv*): i.v. thrombolysis with rtPA
  Interventions: Procedure: Intravenous Thrombolysis
- 2 (L*): intraarterial thrombolysis
  Interventions: Procedure: Intraarterial Thrombolysis

INTERVENTIONS:
Procedure: Intravenous Thrombolysis — i.V. thrombolysis with rtPa
  Groups: 1 1 (Liv*)
Procedure: Intraarterial Thrombolysis — Endovascular treatment with i.a. Urokinase or i.a. rtPA or mechanical recanalization techniques
  Groups: 2 (L*)

SUMMARY:
The clinical and radiological data of patients with an acute ischemic stroke treated with intravenous thrombolysis (IVT) or intraarterial thrombolysis (IAT) in a Swiss stroke unit are assessed in a Swiss Multicenter Thrombolysis Registry. Like in clinical routine, a clinical evaluation takes place in a 3-months follow-up. Furthermore quality of life is assessed with a standardized questionnaire. The aim of the registry is to compare the safety and efficacy of IVT and IAT in patients with acute ischemic stroke. The registry also helps to improve in-hospital-management of stroke patients.

DETAILED DESCRIPTION:
Background: Intravenous thrombolysis (IVT) and intra-arterial thrombolysis (IAT) have been shown to be effective treatments for acute stroke in controlled randomized trials and meta-analyses. However, prospective studies comparing IVT and IAT have not been performed, and it is not known which patients benefit more from IVT or IAT. Non-invasive neurovascular imaging techniques such as magnetic resonance angiography (MRA) or computed tomography angiography (CTA) have the potential to improve patient selection for the optimal mode of thrombolytic therapy and provide data of pre-treatment neurovascular findings of patients treated with IVT. IAT series have identified several prognostic factors for favourable or poor outcome predictors such as vessel recanalization, location of the vascular occlusion or NIHSS at admission. Additional studies have shown that recanalization rates in patients with central ves-sel occlusions such as middle cerebral artery (MCA) main stem or MCA main branch or basilar artery (BA) is higher when treated with IAT compared to IVT. Therefore, the investigators hypothesize that IAT might be more efficacious in these patients.

Objective: Prospective observational multicenter registry with the following aims: To compare the safety and efficacy of IAT and IVT in patients with acute ischemic stroke. To improve safety of IAT and IVT by monitoring the in-hospital management.

Methods: Consecutive patients with acute ischemic stroke who are treated with IVT or IAT within 6 hours of symptom onset in a Swiss stroke unit will be eligible for this registry. Patients are given either intravenous rt-PA or receive IAT such as intra-arterial urokinase, intra-arterial rt-PA or mechanical endovascular recanalization techniques. Patient involvement in the registry shall not influence any treatment decision. Patients will undergo a complete diagnostic work up including a clinical neurological examination using the National Institutes of Health Stroke Scale (NIHSS) score on admission, laboratory examination, brain and neurovascular imaging, echocardiography, 24-hours ECG to determine stroke etiology using the Trial of Org 10172 in Acute Stroke Treatment (TOAST) criteria. The treating physician will initiate secondary prevention of stroke as soon as possible. All patients will be examined by CT and CTA or MRI and MRA on day 1 and in any case of clinical deterioration to exclude intracranial haemorrhage and to assess recanalization of the occluded vessel (using the thrombolysis in myocardial infarction (TIMI) grading system). Clinical outcome will be evaluated on day 1 and at 3 months using the National Institute of Health Stroke Scale (NIHSS) score, modified Rankin Scale score (mRS), Barthel Index (BI), and assessing adverse events and quality of life. The proportion of patients with favourable outcome (mRS 0 to 2) at 3 months after IVT and IAT will serve as the primary outcome measure. In addition, subgroup analyses will be performed stratified by NIHSS, location of vessel occlusion, time to hospital admission and time to treatment. Secondary outcome measures will include quality of life and the proportion of patients with an excellent outcome (mRS 0 or 1) at 3 months, BI 75 to 100 at 3 months, mortality at 3 months, rapid neurological improvement during the first 24 hours, complete or partial recanalization, and symptomatic intracranial haemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Intracranial arterial occlusion confirmed by conventional angiography, MRA or CTA
* National Institute of health Stroke Scale (NIHSS) score ≥ 4 or isolated aphasia or hemianopia
* Time to treatment < 6 hours

Exclusion Criteria

* Intracranial haemorrhage on CT scn or MRI
* History of intracranial haemorrhage or subarachnoid haemorrhage
* Platelet count < 100'000
* International normalized ration (INR) > 1.5
* Partial thromboplastin time (PTT) > 1.5 times the normal value
* Known hereditary of acquired haemorrhagic diathesis
* Pre-existing neurological deficit (mRS>2)
* Previous stroke that might interfere with the neurological assessment (mRS >2)
* Active gastric ulcer
* Major trauma within the preceding 3 months
* Major surgery within the past 4 weeks
* Childbirth within the previous 4 weeks
* Pregnancy
* Uncontrolled hypertension (>185/10 on repeated measures despite antihypertensive medication)
* Severe systemic disease with poor prognosis (e.g. cancer, severe heart failure)
* Intracranial neoplasm
* Combined IVT and IAT
* Combined Intravenous and Ultrasound Thrombolysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute ischemic stroke treated with intravenous or intra-arterial thrombolysis in a Swiss Stroke Unit.
Sampling Method: Non-Probability Sample
Enrollment: 1476 (Actual)
Dates: Start 2007-12; Primary Completion 2015-03 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
overall frequency of favourable clinical outcome (modified Rankin Scale 0 to 2), and unfavourable clinical outcome or death (modified Rankin Scale 3 to 6) | Day 90

SECONDARY OUTCOMES:
subgroup analyses will be performed stratified by NIHSS score | Day 90
Excellent functional clinical outcome (modified Rankin Scale 0 or 1) and quality of life (measured by EuroQol and Stroke specific Quality of Life Scale) | Day 90
All causes of mortality | Day 90
Proportion of patients with rapid neurological improvement (more than 4 points on the NIHSS) during the first 24 hours after thrombolysis. | Day 1
Complete or partial recanalization of the occluded artery (TIMI grade 2 or 3) assessed by CTA or MRA. | Day 1
Symptomatic intracranial haemorrhages up to 24 hours after thrombolysis defined as homogeneous areas of haemorrhage, with or without mass effect or intraventricular extension with neurological deterioration | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Marcel Arnold, MD Prof., Principal Investigator — Dep. of Neurology, Bern University Hospital, Switzerland; Krassen Nedeltechev, MD Prof., Principal Investigator — Kantonsspital Aarau, Switzerland
Locations (1):
- Dep. of Neurology, Bern University Hospital, Bern, Switzerland